CLINICAL TRIAL: NCT01043146
Title: A Single-Blind Placebo-Controlled Dose Escalating Safety and Pharmacokinetic Study of an Acute Intravenous Administration of Cor-1, An Anti-ß1 Receptor Antibody Cyclopeptide, in Five Different Strengths in Healthy Male Volunteers
Brief Title: Safety, Pharmacokinetic and Pharmacodynamic Study of COR-1, an Anti-ß1 Receptor Antibody Cyclopeptide
Acronym: COR-1-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corimmun GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COR-1-01; EudraCT2008-007745-31 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Results first posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-03

CONDITIONS: Heart Failure
Keywords: anti-beta1 adrenergic receptor; autoantibody; cyclic peptide; heart failure
MeSH Terms: conditions — Heart Failure | interventions — Peptides, Cyclic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- COR-1 (Active Comparator): single intravenous administration of 10, 40, 80, 160 or 240 mg of COR-1
  Interventions: Drug: COR-1
- placebo (Placebo Comparator): intravenous 0.9 % NaCl
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: COR-1 — single intravenous administration of 10, 40, 80, 160 or 240 mg of COR-1
  Other Names: cyclic peptide
  Arms: COR-1
Drug: placebo — intravenous 0.9 % NaCl
  Arms: placebo

SUMMARY:
Primary Trial objectives:

To evaluate the pharmacokinetics and -dynamics of five strengths of COR-1 (10, 40, 80, 160, 240 mg) in 50 healthy, male volunteers after single intravenous administration (8 subjects on verum per dose level, 10 subjects receiving placebo)

Secondary objectives:

To evaluate safety and tolerability by using adverse events (AEs) and vital signs

DETAILED DESCRIPTION:
Primary Trial objective:

To evaluate the pharmacokinetics and -dynamics of five strengths of COR-1 (10, 40, 80, 160, 240 mg) in healthy, male volunteers after single intravenous administration

Secondary objectives:

To evaluate safety and tolerability by using adverse events (AEs), vital signs including blood pressure/pulse rate (BP/PR), electrocardiographic examinations (12 lead ECG), evaluation of antibody titer and safety laboratory tests (biochemistry, hematology, coagulation, urinalysis)

Methodology:

Mono-center, single-blind, dose escalating study with five dose levels (8 subjects on verum per dose level, 2 subjects receiving placebo) in a total of 50 volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male Caucasians between 18 and 45 years of age, inclusive
* Normotensive subjects (systolic BP <140 mmHg and diastolic BP <90 mmHg)
* Body mass index (BMI) 19-27, minimal weight 60 kg
* Negative results in HIV antibody, HBs antigen (HBsAg) and HCV tests, and negative result in anti-ß1-receptor-autoantibody screening
* Signed Informed Consent Form
* Normal or clinically irrelevant laboratory findings

Exclusion Criteria:

* Autoimmune disorders
* Kidney diseases
* Liver diseases, liver function impairments

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mariola Lappo, MD, Principal Investigator — ABX CRO
Locations (1):
- ABX-CRO, Görlitz, Saxony, Germany

REFERENCES:
- [Derived] Munch G, Boivin-Jahns V, Holthoff HP, Adler K, Lappo M, Truol S, Degen H, Steiger N, Lohse MJ, Jahns R, Ungerer M. Administration of the cyclic peptide COR-1 in humans (phase I study): ex vivo measurements of anti-beta1-adrenergic receptor antibody neutralization and of immune parameters. Eur J Heart Fail. 2012 Nov;14(11):1230-9. doi: 10.1093/eurjhf/hfs118. Epub 2012 Sep 11. PMID 22968742

RESULTS

PARTICIPANT FLOW:
Groups:
- 10 mg COR-1; 40 mg COR-1; 80 mg COR-1; 160 mg COR-1; 240 mg COR-1: single intravenous administration
Period: Overall Study
Arm/Group | Placebo | 10 mg COR-1 | 40 mg COR-1 | 80 mg COR-1 | 160 mg COR-1 | 240 mg COR-1
Started | 10 | 8 | 8 | 8 | 8 | 8
Completed | 10 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg COR-1 | 40 mg COR-1 | 80 mg COR-1 | 160 mg COR-1 | 240 mg COR-1 | Total
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 8 | 8 | 8 | 8 | 8 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.1 (8.61) | 32.5 (7.09) | 33.1 (8.94) | 31.9 (7.77) | 30.1 (8.66) | 27.5 (8.35) | 31.6 (8.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 10 | 8 | 8 | 8 | 8 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Reporting Adverse Events (AEs)
Description: To assess the safety and tolerability of COR-1.
Time Frame: 45 days
Measure: Number; unit: Participants
Arm/Group | Placebo | 10 mg COR-1 | 40 mg COR-1 | 80 mg COR-1 | 160 mg COR-1 | 240 mg COR-1
Number analyzed (Participants) | 10 | 8 | 8 | 8 | 8 | 8
Participants
  AE | 0 | 0 | 3 | 0 | 0 | 0
  SAE | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Placebo | 10 mg COR-1 | 40 mg COR-1 | 80 mg COR-1 | 160 mg COR-1 | 240 mg COR-1
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 0/8 | 0/8 | 0/8 | 1/8
Other Adverse Events (participants affected / at risk) | 0/10 | 0/8 | 3/8 | 0/8 | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 10 mg COR-1 (N=8) | 40 mg COR-1 (N=8) | 80 mg COR-1 (N=8) | 160 mg COR-1 (N=8) | 240 mg COR-1 (N=8)
not drug-related traumatic injury (achilles tendon) during sledging 8600 half-lives post drug admin. (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Injury by sheet metal used for tobogganing 18 days after drug administration. Hospitalisation for 3 days (2 nights). Plastic reconstruction of the Achilles tendon, antibiotic treatment and wound dressing. Ambulatory follow up 31 days later.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=10) | 10 mg COR-1 (N=8) | 40 mg COR-1 (N=8) | 80 mg COR-1 (N=8) | 160 mg COR-1 (N=8) | 240 mg COR-1 (N=8)
feeling of cold at infusion site when drug was added to cold saline solution (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Caused by cold temperature of infusion solution. The event never reoccurred when solution was equilibrated to room temperature prior to injection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can discuss and publish trial results upon review of results communication by the sponsor. The sponsor can require changes to the communication.